CLINICAL TRIAL: NCT06974903
Title: A RetrospectiVe ObservatIoNal Study of a CurrEnt Status and Its Management of GERD (GastroEsophageal Reflux Disease) in General HOspitals in Korea
Brief Title: Retrospective Observational Study on GERD Management in General Hospitals in Korea
Acronym: VINCERO
Status: Completed | Type: Observational
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: D999_02GERD2003
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: GastroEsophageal Reflux Disease; GERD; Korean patients; Observational study; RetrospectiVe Observational study
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A RetrospectiVe ObservatIoNal Study of a CurrEnt Status and its Management of GERD (GastroEsophageal Reflux Disease) in General HOspitals in Korea

DETAILED DESCRIPTION:
This study is designed as a multicenter, retrospective observational study. After signing a contract with the research institution or investigator, patients who meet the inclusion/exclusion criteria in the study protocol will be enrolled. The registration of patients at each research site will be carried out in order based on the most recent visit date (or GERD diagnosis date) as of January 1, 2018. Data from the study subjects will be collected by reviewing medical records from January 1, 2018, to August 31, 2020. These data will be recorded in the eCRF through interviews, examinations, and tests performed under the investigator's judgment during routine clinical practice within this period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years or older as of the date of their first visit.
2. Patients who visited domestic general hospitals (secondary and tertiary healthcare institutions) at least twice between January 1, 2018, and August 31, 2020, for the diagnosis or treatment of GERD.

Exclusion Criteria:

1. Patients with no GERD treatment information recorded in the medical records, even once.
2. Patients deemed inappropriate for participation by the investigator (e.g., when the overall GERD diagnosis/treatment information is missing from the medical records).

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Gastroesophageal Reflux Disease(GERD)
Sampling Method: Probability Sample
Enrollment: 13750 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of Incidence of Adverse events following the administration of GERD treatment medications | From enrollment to 2 years and 7 months after registration
  the safety assessment of all adverse events occurring after GERD medication treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Hospital, Seoul, Seongdong-gu, South Korea